CLINICAL TRIAL: NCT05457699
Title: Ablative Radiotherapy to Consolidate Maximal Systemic Response in Metastatic Prostate Cancer (ANCHOR-Prostate)
Acronym: ANCHORProstate
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.115
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR consolidation (Experimental)
  Interventions: Radiation: SABR
- Control - no SABR consolidation (Active Comparator)
  Interventions: Other: no RT

INTERVENTIONS:
Radiation: SABR — SBAR to PSMA-PET visible disease at maximal systemic therapy response.
  Arms: SABR consolidation
Other: no RT — no SABR, continued systemic therapy per SOC
  Arms: Control - no SABR consolidation

SUMMARY:
A phase IIR cmRCT trial companion to PERa registry, investigating the merit of SABR consolidation in men with metastatic prostate cancer. 80 patients will be randomly selected to be offered experimental SABR based on PSMA-PET detected disease after maximal systemic response. The primary endpoint is the rate of FFS at 1 year. Patients will be stratified according to hormone sensitive vs resistant disease prior to randomisation.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Enrolled in PERa (CHUM CER 17.032) and randomly selected for AnChoR-Prostate.

3.1.2 Diagnosis of metastatic prostate cancer having achieved maximum PSA response to SOC systemic therapy defined as two consecutive stable PSA within 6 months of regimen start. Stable PSA is defined as non- progressing (<25% rise from nadir, per PCWG3 guidelines).

3.1.3 ECOG 0-2 3.1.4 PSA > 0.2 ng/mL 3.1.5 1-5 sites of PSMA-PET avid disease amenable to SABR.

Exclusion Criteria:

* none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
FFS | 1 year
  FFS is defined as time from randomization to the first of the following events: PSA progression, radiographic or clinical progression.

SECONDARY OUTCOMES:
HRQoL | 5 years
Toxicity | 5 years
  CTCAEv5, incidence rate
Time to progression | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CRCHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided